CLINICAL TRIAL: NCT05309941
Title: The Effects of External Cues Versus Internal Cues Messaging on Heart Rate Variability and Affect
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Responsible Party: Principal Investigator, Carly R Pacanowski, Assistant Professor, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: 1846581
Record Dates: First submitted 2022-02-10; First posted 2022-04-04 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Dietetics; Diet, Healthy; Nutrition Therapy; Affect; Autonomic Nervous System
Keywords: nutrition messaging; nutrition education; Intuitive Eating

STUDY DESIGN:
Intervention Model Description: Participants attend a single study visit and are randomized to view one of two nutrition education videos.
Who Masked: Participant
Masking Description: The participants are not aware of the condition they are assigned to.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Internal Cues Messaging (Experimental): Participants will view a five-minute video focusing on intuitive eating principles.
  Interventions: Other: Internal Cues Nutrition Messaging
- External Cues Messaging (Active Comparator): Participants will view a five-minute video focusing on traditional nutrition education principles.
  Interventions: Other: External Cues Nutrition Messaging

INTERVENTIONS:
Other: Internal Cues Nutrition Messaging — Participants will view a 5 minute nutrition education video focused on intuitive eating principles.
  Arms: Internal Cues Messaging
Other: External Cues Nutrition Messaging — Participants will view a 5 minute nutrition education video focused on traditional nutrition education principles such as label reading.
  Arms: External Cues Messaging

SUMMARY:
This randomized controlled trial will assess the effects of External Cues focused messaging (i.e., government recommendations of MyPlate) compared to Internal Cues focused messaging (i.e., intuitive eating). The investigators will collect data on within-person changes in psychological (e.g. affect) and physiological (e.g. heart rate variability) outcomes in female college students.

Participants will be randomly assigned to one of two study conditions. In condition one, participants will view a five-minute video focusing on traditional nutrition education principles. In condition two, participants will view a five-minute video focusing on intuitive eating principles.

ELIGIBILITY:
Inclusion Criteria:

* 18-29 years old
* identify as female
* college student

Exclusion Criteria:

* outside of the age range of 18-29 years
* do not self-identify as female
* not able to attend an in-person study visit at the University of Delaware

Ages: 18 Years to 29 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Individuals who identify as female are eligible to participate.
Enrollment: 300 (Actual)
Dates: Start 2022-01-20 (Actual); Primary Completion 2022-12-20 (Actual); Study Completion 2022-12-20 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) | HRV will be measured during a 3-minute baseline period and while watching a 5-minute intervention video.
  Heart rate variability measures the variation in time between each heartbeat. This will be measured using Firstbeat Electrocardiograms (ECGs) that participants will attach to their chest using two electrodes.
Change in Affect | The PANAS is administered before and immediately after viewing the video.
  Affect will be assessed using the Positive and Negative Affect Schedule (PANAS), an instrument that asks participants to rank the extent to which they are feeling each of 20 different emotions on a scale of 1-5. The PANAS produces a score from 10-50 for each Positive Affect and Negative Affect, with higher scores indicating higher levels of these states.

CONTACTS AND LOCATIONS:
Overall Officials: Carly R Pacanowski, PhD RD, Principal Investigator — University of Delaware; Christine Skubisz, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

IPD SHARING:
Plan to Share IPD: Yes
Dataset
Supporting Information: Study Protocol, ICF

REFERENCES:
- [Derived] Pacanowski CR, Vizthum D, Cash H, Katcher JA, Skubisz C. A weight-centric health message elicits higher body shame in those at risk for eating disorders. Appl Psychol Health Well Being. 2025 Aug;17(4):e70061. doi: 10.1111/aphw.70061. PMID 40781768